CLINICAL TRIAL: NCT05968391
Title: Comparison of Acetoacetate and Acetate Kidney Uptake in Patients With Chronic Kidney Failure Measured by Positron Emission Tomography : the RENO-TEP Project
Brief Title: Acetoacetate and Acetate Metabolism in Patients With Chronic Kidney Failure.(RENO-TEP)
Acronym: RENO-TEP
Status: Recruiting | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Collaborators: Nestle Health Science (Industry)
Responsible Party: Sponsor
Other Study IDs: 2024-5157
Record Dates: First submitted 2023-07-20; First posted 2023-08-01 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Kidney Failure, Chronic
Keywords: ketone; acetoacetate; acetate
MeSH Terms: conditions — Kidney Failure, Chronic; Ketosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic kidney failure: No interventions for the purpose of the study. They will simply undergo two PET scans consecutively
  Interventions: Radiation: PET scan metabolic day

INTERVENTIONS:
Radiation: PET scan metabolic day — 11C-Acetate and 11C-Acetoacetate PET scans

SUMMARY:
The objective of this study is to nake a comparison between 11c-acetate and 11c-acetoacetate kidney uptake in chronic kidney failure patients.

DETAILED DESCRIPTION:
Chronic kidney failure patients will be ask to perform two positron emission tomography scan during the same day. One, with a 11C-Acetate Tracer and the other with 11C-Acetoacetate. The results will allow to determine the difference between the two tracers and will ultimately be compared with precedent results of healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.5 and 40
* Kidney failure if GFR betweem 30 and 60 mL/min/1.73m2
* Stable medication for at least 4 weeks

Exclusion Criteria:

1. Receive cytotoxic therapy for primary or secondary kidney disease within 6 months prior to enrollment
2. Organ Transplant History
3. Class IV congestive heart failure (New York Heart Association)
4. Myocardial infarction, unstable angina, stroke or transient ischemic attack within 12 weeks prior to enrollment
5. Coronary revascularization (percutaneous coronary intervention or arterial bypass) or valve repair/replacement within 12 weeks of enrollment or is scheduled to undergo one of these procedures within 4 weeks of enrollment
6. Any condition outside the realm of renal and cardiovascular disease, such as, but not limited to, malignancy, with a life expectancy of less than 2 years in the clinical judgment of the investigator
7. Active malignancy requiring treatment at Visit 1 (except successfully treated basal or squamous cell carcinoma).
8. Hepatic impairment (aspartate transaminase or alanine transaminase >3x upper limit of normal; or total bilirubin >2x upper limit of normal at time of enrollment
9. Pregnancy or lactation
10. Adherence to a ketogenic diet, consumption of ketogenic products or supplements or intermittent fasting or other diet or supplements that may significantly increase ketones in the past two months.
11. Daily alcohol consumption >2 servings per day
12. Participation in other interventional research projects concurrently or participation in other PET research projects in the last year, which exceeds the recommended limits
13. Inability to lie still in supine position;
14. Medical fluid restriction limiting fluid intake for the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with kidney failure
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Mean in kidney acetate uptake | 30 minutes
  Kidney acetate uptake measured by pet scan
Mean in kidney acetoacetate uptake | 30 minutes
  Kidney acetoacetate uptake measured by pet scan
Mean in kidney acetoacetate metabolism | 30 minutes
  Kidney acetoacetate metabolism measured by pet scan
Mean in kidney acetate metabolism | 30 minutes
  Kidney acetate metabolism measured by pet scan

SECONDARY OUTCOMES:
Mean in heart ejection fraction | 30 minutes
  Ejection fraction measured by pet scan

CONTACTS AND LOCATIONS:
Overall Officials: Mélanie Godin, MD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre de recherche sur le vieillissement, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No